CLINICAL TRIAL: NCT04648527
Title: Prospective Study of Arthroscopic Diagnosis and Treatment of the Isolated Dorsal Wrist Syndrome in Patients With Hypertrophy of the Dorsal Synovial
Brief Title: Arthroscopic Diagnosis and Treatment of Dorsal Wrist Syndrome in Patients With Synovial Hypertrophy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Consorci Sanitari Integral (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20/31
Record Dates: First submitted 2020-11-18; First posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Synovial Hypertrophy Hand (Diagnosis)
Keywords: wrist; arthroscopy; synovectomy
MeSH Terms: conditions — Disease | interventions — Electrocoagulation

STUDY DESIGN:
Intervention Model Description: Prospective before-and-after study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: arthroscopic synovectomy and thermocoagulation — An diagnostic arthroscopy and an arthroscopic synovectomy and thermocoagulation of the dorsal hypertrophic synovial will be performed

SUMMARY:
The objective of the study is to evaluate de results of the arthroscopic diagnose and arthroscopic treatment of the dorsal wrist pain syndrome associated with dorsal synovial hypertrophy.

It is a prospective study of 25 consecutive patients with the diagnosis of dorsal wrist radiographies and MRI) have discarded other concomitant pathologies. After being refractory to the conservative measures consisting in physiotherapy for at least 3 months, a wrist arthroscopy will be performed with diagnostic and treatment objectives. All these procedures will be performed by the same surgical team. Only will be included those patients whose diagnostic arthroscopy show absence of other concomitant lesions as scapho-lunate or luno-triquetral tears, triangular fibrocartilage injuries, chondral injuries, fractures, arthritis or other injuries that will be considered as exclusion criteria. In those cases where a hypertrophy of the dorsal synovial is confirmed, an arthroscopic synovectomy and radiofrequency thermocoagulation of the hypertrophic synovial will be performed. The standard radiocarpal portals for wrist arthroscopy will be performed: 3-4 portal and 6-R portal.

The pain syndrome described as dorsal localized wrist pain, especially reproductible in hyperextension and axial load of the wrist and in whom the complementary tests (plain The following data will be reviewed and analyzed: age, sex, right/left wrist, right/left-handed, anamnesis, physical exam, MRI findings, arthroscopic diagnosis and functional outcome through Mayo score as a main viable and also, VAS(visual analogue scale for pain), DASH score, grip strength measured with jamar dynamometer and articular balance. All these parameters will be registered pre-surgery and post-surgery at 6 weeks, 3 months and 12 months of the follow-up and at the end of follow-up. The minimum follow-up will be at least of 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women
2. Age 18-65 years old, both included
3. Diagnose of primary dorsal wrist syndrome, defined as:

   3.1 Radiocarpal dorsal focal pain 3.2 Pain increases in hyperextension of the wrist and in axial load 3.3 X-rays and MRI without significant findings 3.4 Watson test, extension finger test, Kleinman shuck test, distal radio-ulnar ballottement test, fovea sign all of them negatives and absence of tenosynovitis of the extensor tendons.
4. Refractory to conservative treatment consisting in at least 3 months of physical therapy.
5. Presence of a hypertrophy of the dorsal synovial of the wrist diagnosed through direct visualization in wrist arthroscopy.
6. Other diagnoses excluded through wrist arthroscopy

Exclusion Criteria:

1. Hand or wrist fractures
2. Arthritis
3. Carpal boss
4. Scapho-lunate ligament tears
5. Luno-triquetral ligament tears
6. Triangular fibrocartilage tears
7. Bone necrosis
8. Systemic arthritis as rheumatoid arthritis, psoriasic arthritis, gouty arthritis, etc.)
9. Dorsal or volar ganglions
10. Distal radio-ulnar joint injury or instability
11. Hand or wrist infections or tumors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the Mayo wrist score | Before intervention, 3 months after intervention, 6 months after intervention, 12 months after intervention
  Assessment of the changes of Mayo score, before the intervention and at 3 months, 6 months and 12 months after the intervention. The Mayo wrist score ranges from 0 to 100 with a score of 0 indicating a worse wrist condition and 100 indicating a better wrist condition.

CONTACTS AND LOCATIONS:
Overall Officials: Camila Chanes Puiggrós, MD, Principal Investigator — Hospital Dos de Maig, Consorci Sanitari Integral
Locations (1):
- Hospital Dos de Maig, Consorci Sanitari Integral, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No